CLINICAL TRIAL: NCT03057301
Title: Assessment of Home Tonometry in Glaucoma
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC16040
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Glaucoma; Intraocular Pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: iCare home tonometer — All subjects will be taught to use the home care tonometer.

SUMMARY:
Worldwide, glaucoma is the most common cause of irreversible blindness. The major risk factor is raised pressure within the eye (intraocular pressure, IOP). IOP is typically measured using Goldman applanation tonometry (GAT). This involves instilling anaesthetic eye drops and using a probe to contact the cornea and obtain a pressure measurement. A major disadvantage of GAT is that only limited numbers of pressure measurements can be obtained, whereas IOP is known to vary throughout the day and in ¾ of people is highest during the night. The result is that clinicians have poor understanding of patient's 24 hour IOPs and the effect that this might have on their glaucoma. This is a serious limitation as the treatment of glaucoma depends on lowering IOP.

Recently a new device has become available, designed specifically for home IOP monitoring. The iCare HOME tonometer is a CE marked commercial device (http://www.icaretonometer.com/products/icare-home-tonometer/) that can be used to gain insight into 24-hour IOP fluctuations. The investigators wish to determine the feasibility of home IOP monitoring using this device. The iCare HOME tonometer depends on the patient performing self-tonometry. Testing one's own IOP may be technically difficult and it is likely that large numbers of patients will struggle with this.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma
* At least 4 previous visual field tests (to enable rate of change to be calculated).
* Age 16 years and above
* Age less than 100

Exclusion Criteria:

* Corneal disease (potentially affects pressure measurements)
* Neovascular glaucoma
* Uveitis
* Secondary glaucomas
* Inability to give informed consent.
* Less than 16 years of age.
* Pregnancy.
* Unable to hold iCare HOME® tonometer due to upper limb weakness or disability.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with glaucoma attending a university hospital glaucoma clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Whether or not the subject is deemed successful in using the home tonometer | On baseline visit
  Strict success = intraocular pressure within 5mmHg of that obtained by technician

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Tatham, FRCOphth, Principal Investigator — NHS Lothian
Locations (1):
- Princess Alexandra Eye Pavilion, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No